CLINICAL TRIAL: NCT04830124
Title: A Phase 2, Open-Label, Multicenter, Cohort Study of Nemvaleukin Alfa (ALKS 4230) Monotherapy and in Combination With Pembrolizumab in Patients With Advanced Cutaneous Melanoma or Advanced Mucosal Melanoma - ARTISTRY-6
Brief Title: Nemvaleukin Alfa Monotherapy and in Combination With Pembrolizumab in Patients With Advanced Cutaneous or Mucosal Melanoma - ARTISTRY-6
Acronym: ARTISTRY-6
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated due to business and strategic decision.
Sponsor: Mural Oncology, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALKS 4230-006
Record Dates: First submitted 2021-04-01; First posted 2021-04-02 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Cutaneous Melanoma; Mucosal Melanoma
Keywords: ALKS 4230; Melanoma; Immunotherapy; Nemvaleukin alfa; IL-2; Interlukin-2; Oncology; Cytokine; Nemvaleukin; Mural Oncology; Pembrolizumab
MeSH Terms: conditions — Melanoma; Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Advanced Cutaneous Melanoma Subcutaneous Dosing (Cohort 1) (Experimental): Patients with unresectable and/or metastatic cutaneous melanoma
  Interventions: Drug: Nemvaleukin Alfa Subcutaneous
- Advanced mucosal melanoma with IV Dosing (Cohort 2) (Experimental): Patients with unresectable and/or metastatic mucosal melanoma
  Interventions: Drug: Nemvaleukin Alfa Intravenous
- Advanced Cutaneous Melanoma with Less Frequent IV Dosing (Cohort 3) (Experimental): Patients with unresectable and/or metastatic cutaneous melanoma
  Interventions: Drug: Nemvaleukin Alfa Intravenous Less Frequent Dosing
- Advanced Cutaneous Melanoma with Less Frequent IV Nemvaleukin Dosing + Pembrolizumab (Cohort 4) (Experimental): Patients with unresectable and/or metastatic cutaneous melanoma. Patients must not have received prior systemic anticancer therapy for unresectable or metastatic melanoma. Prior adjuvant and/or neoadjuvant PD-[L]1 treatments are allowed if there is at least 6 months between the last dose and date of recurrence.
  Interventions: Drug: Nemvaleukin Alfa Intravenous Less Frequent Dosing; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Nemvaleukin Alfa Subcutaneous — Subcutaneous injection of nemvaleukin every 7 days
  Other Names: ALKS 4230 Subcutaneous
  Arms: Advanced Cutaneous Melanoma Subcutaneous Dosing (Cohort 1)
Drug: Nemvaleukin Alfa Intravenous — Intravenous (IV) infusion over 30 minutes given daily for 5 consecutive days
  Other Names: ALKS 4230 Intravenous
  Arms: Advanced mucosal melanoma with IV Dosing (Cohort 2)
Drug: Nemvaleukin Alfa Intravenous Less Frequent Dosing — Intravenous (IV) infusion over 30 minutes twice every 21 days (Day 1 and Day 8 dosing of a 21 day cycle)
  Other Names: ALKS 4230 Intravenous
  Arms: Advanced Cutaneous Melanoma with Less Frequent IV Dosing (Cohort 3); Advanced Cutaneous Melanoma with Less Frequent IV Nemvaleukin Dosing + Pembrolizumab (Cohort 4)
Drug: Pembrolizumab — Cohort 4 only: 200mg IV pembrolizumab on Day 1 of a 21-day cycle
  Other Names: Keytruda
  Arms: Advanced Cutaneous Melanoma with Less Frequent IV Nemvaleukin Dosing + Pembrolizumab (Cohort 4)

SUMMARY:
This study observes the antitumor activity, safety, tolerability, PK, and pharmacodynamics in patients with inoperable and/or metastatic melanoma

ELIGIBILITY:
Inclusion Criteria:

* The patient must have the following tumor types:

Cohort 1: Patient has unresectable and/or metastatic cutaneous melanoma. No more than 5 patients with acral melanoma may enroll in this cohort.

Cohort 2: Patient has unresectable and/or metastatic mucosal melanoma.

Cohort 3: Patient has unresectable and/or metastatic cutaneous melanoma. Patients with acral melanoma may not enroll in this cohort.

Cohort 4: Patient has unresectable and/or metastatic cutaneous melanoma. No patients with mucosal or acral melanoma may enroll in this cohort.

- The patient must have received previous treatment as follows: Cohorts 1 and 2: Patient has received anti-PD-[L]1 therapy with or without anti-CTLA-4 therapy, and less than or equal to one other prior regimen of systemic anti-neoplastic therapy (eg, targeted therapy, chemotherapy). Previous adjuvant and/or neoadjuvant therapy counts as one prior regimen. Patients have experienced objective response (partial response [PR] or CR; by RECIST 1.1 or iRECIST) or stable disease (SD; by RECIST 1.1 or iRECIST) as best overall response (BOR) to anti-PD-[L]1 therapy. Patients with confirmed progressive disease (by RECIST 1.1 or iRECIST) as best response may be included, if they received anti-PD-[L]1 therapy for a minimum of 12 weeks (eg, from first dose to last dose). Patients with BRAF mutations may or may not have received prior targeted therapy.

Cohort 3: Patients who have received anti-PD-[L]1 therapy with or without anti-CTLA-4 therapy or anti-lymphocyte-activation gene 3 (LAG-3) therapy, and ≤1 other prior regimen of systemic anti-neoplastic therapy (eg, targeted therapy, chemotherapy). Previous adjuvant and/or neoadjuvant therapy counts as 1 prior regimen. Patients must have experienced objective response (PR or CR by RECIST 1.1 or iRECIST) or stable disease (by RECIST 1.1 or iRECIST) as BOR to anti PD-[L]1 therapy. Patients with confirmed progressive disease (by RECIST 1.1 or iRECIST) as best response may be included, if they received anti-PD-[L]1 therapy for ≥12 weeks (from first dose to last dose). Patients with BRAF mutations may or may not have received prior targeted therapy.

Cohort 4: Patients must not have received prior systemic anticancer therapy for unresectable or metastatic melanoma. Prior adjuvant and/or neoadjuvant PD-[L]1 treatments are allowed if there is at least 6 months between the last dose and date of recurrence.

Cohorts 1, 2, and 3 - Patients who have received prior treatment with talimogene laherparepvec (TVEC) are allowed to enroll provided that last exposure to TVEC was ≥28 days prior to first exposure to nemvaleukin and that all injection-site reactions to TVEC have resolved. TVEC shall not be considered a prior regimen of systemic anti-neoplastic therapy, nor shall it be considered a systemic immunomodulatory agent.

* Patients must have disease that is measurable based on RECIST 1.1., that has not recently been irradiated or used to collect a biopsy.
* Cohorts 1 and 2 (required), Cohort 3 (optional), Cohort 4 (may be required, otherwise optional). Patient is willing to undergo a pretreatment tumor biopsy or provide qualifying archival tumor tissue.

Cohort 4 - Patients are required to have known tumor PD-[L]1 status determined by local testing using an approved assay. PD-[L]1 testing performed prior to enrolling on the study is acceptable if there was no intervening systemic anti-cancer therapy, and archival tissue may be used for testing provided the biopsy is ≤3 months old.

* Patient has an Eastern Cooperative Oncology Group (ECOG) status of 0 or 1 and an estimated life expectancy of ≥3 months.
* Additional criteria may apply.

Exclusion Criteria:

* Patient has uveal melanoma (all cohorts) or acral melanoma (Cohort 2, Cohort 3 and Cohort 4).
* Patient has received prior interleukin (IL)-2-based or IL-15-based cytokine therapy; patient has had exposure, including intralesional, to IL-12 or analogs thereof.
* Patient requires systemic corticosteroids (>10 mg of prednisone daily, or equivalent) however, replacement doses, topical, ophthalmologic, and inhalational steroids are permitted.
* Patient has undergone prior solid organ and/or non-autologous hematopoietic stem cell or bone marrow transplant.
* Patient is currently pregnant, breastfeeding, or is planning to become pregnant or to begin breastfeeding during the study period or within 30 days (Cohorts 1,2, and 3) or 120 days (Cohort 4) after last study drug administration.
* Patients with active or symptomatic central nervous system metastases unless the metastases have been treated by surgery and/or radiation therapy and/or gamma knife, the subject has been tapered to a dose of 10 mg of prednisone (or equivalent) or less of corticosteroids for at least 2 weeks before the first dose, and the subject is neurologically stable. Patients with leptomeningeal disease are excluded.
* Patient has known or suspected hypersensitivity to any components of nemvaleukin (all cohorts) or to pembrolizumab (cohort 4 only).
* Patients with an uncontrollable bleeding disorder.
* Patient has QT interval corrected by the Fridericia Correction Formula values of >470 msec (in females) or >450 msec (in males); patient who is known to have congenital prolonged QT syndromes; or patient who is on medications known to cause prolonged QT interval on ECG.
* Patient has developed Grade ≥3 immune-related AEs (irAEs) while on prior immunotherapy, (eg, pneumonitis and nephritis) and has not recovered to ≤Grade 1 and/or are on systemic steroids within 14 days of first dose of study drug.
* Patients who have previously discontinued immunotherapy due to immune-related adverse event (irAEs) will be excluded.
* Cohort 4 only: Patient has a history of (noninfectious) pneumonitis that required steroids or has current pneumonitis.
* Additional criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2021-09-27 (Actual); Primary Completion 2025-05-08 (Actual); Study Completion 2025-05-08 (Actual)

PRIMARY OUTCOMES:
Centrally-assessed overall response rate (ORR) (Cohort 1 and 2) | Assessed up to 2 years from the first dose
  * ORR is defined as the number of patients exhibiting a complete response (CR) or partial response (PR) divided by the number of patients who received the study drug
  * Response will be based on RECIST v1.1 criteria
Investigator-assessed overall response rate (ORR) (Cohort 3 and 4) | Assessed up to 2 years from the first dose
  ORR is defined as the number of patients exhibiting a complete response (CR) or partial response (PR) divided by the number of patients who received the study drug

SECONDARY OUTCOMES:
Centrally-assessed duration of response (DOR) (Cohort 1 and 2) | Assessed up to 2 years from the first dose
  -DOR is defined as the time from the first documentation of complete or partial response to the first documentation of either objective tumor progression or death
Investigator-assessed duration of response (DOR) (Cohort 3 and 4) | Assessed up to 2 years from the first dose
  -DOR is defined as the time from the first documentation of complete or partial response to the first documentation of either objective tumor progression or death
Centrally-assessed progression free survival (PFS) (Cohort 1 and 2) | Assessed up to 2 years from the first dose
  -PFS is defined as the time from each respective patient's first dose of nemvaleukin to either the first documentation of objective tumor progression or death
Investigator-assessed progression free survival (PFS) (Cohort 3 and 4) | Assessed up to 2 years from the first dose
  -PFS is defined as the time from each respective patient's first dose of nemvaleukin to either the first documentation of objective tumor progression or death
Centrally-assessed disease control rate (DCR) (Cohort 1 and 2) | Assessed up to 2 years from the first dose
  -DCR is defined as the proportion of patients with objective evidence of complete response, partial response, or stable disease on 2 consecutive protocol-required disease assessments
Investigator-assessed disease control rate (DCR) (Cohort 3 and 4) | Assessed up to 2 years from the first dose
  -DCR is defined as the proportion of patients with objective evidence of complete response, partial response, or stable disease on 2 consecutive protocol-required disease assessments
Centrally-assessed time to response (TTR) (Cohort 1 and 2) | Assessed up to 2 years from the first dose
  -TTR is defined as the time from patient's first dose of nemvaleukin to the first documentation of complete response or partial response
Investigator-assessed time to response (TTR) (Cohort 3 and 4) | Assessed up to 2 years from the first dose
  -TTR is defined as the time from patient's first dose of nemvaleukin to the first documentation of complete response or partial response
Incidence of treatment-emergent adverse events (All cohorts) | Assessed up to 2 years from the first dose
Investigator-assessed overall response rate (ORR) (Cohort 1 and 2) | Assessed up to 2 years from the first dose
  ORR is defined as the number of patients exhibiting a complete response (CR) or partial response (PR) divided by the number of patients who received the study drug
Investigator-assessed immune overall response rate (iORR) (All cohorts) | Assessed up to 2 years from the first dose
  -iORR is defined as the number of patients exhibiting a complete response (CR) or partial response (PR) divided by the number of patients who received the study drug.
Investigator-assessed immune duration of response (iDOR) (All cohorts) | Assessed up to 2 years from the first dose
  -iDOR is defined as the time from the first documentation of complete or partial response to the first documentation of either objective tumor progression or death
Investigator-assessed immune progression free survival (iPFS) (All cohorts) | Assessed up to 2 years from the first dose
  -iPFS is defined as the time from each respective patient's first dose of nemvaleukin to either the first documentation of objective tumor progression or death
Investigator-assessed immune disease control rate (iDCR) (All cohorts) | Assessed up to 2 years from the first dose
  -iDCR is defined as the proportion of patients with objective evidence of complete response, partial response, or stable disease on 2 consecutive protocol-required disease assessments
Investigator-assessed immune time to response (iTTR) (All cohorts) | Assessed up to 2 years from the first dose
  -iTTR is defined as the time from patient's first dose of nemvaleukin to the first documentation of complete or partial response

CONTACTS AND LOCATIONS:
Overall Officials: Mural Oncology Medical Monitor, Study Director — Mural Oncology
Locations (41):
- United States (10):
  - UC San Diego Moores Cancer Center, La Jolla, California
  - The Angeles Clinic and Research Institute, Los Angeles, California
  - Mayo Clinic, Jacksonville, Florida
  - Orlando Health, Inc, Orlando, Florida
  - Norton Cancer Center, Louisville, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - NYU Laura and Isaac Perimutter Cancer Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - UT Southwestern Medical Center of Dallas, Dallas, Texas
- Australia (3):
  - Calvary Mater Newcastle, Waratah, New South Wales
  - John Flynn Private Hospital, Tugun, Queensland
  - The Queen Elizabeth Hospital, Woodville
- Canada (3):
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Centre Hospitalier de l'Universite de Montreal (CHUM), Montreal, Quebec
  - McGill University Health Center (MUHC), Montreal, Quebec
- Italy (6):
  - Istituto Tumori Giovanni Paolo II IRCCS Ospedale Oncologico Bari, Bari
  - Fondazione IRCC Istituto Nazionale dei Tumori, Milan
  - Veneto Oncology Institute, Padua
  - Ospedale S. Maria della Misericordia, Perugia
  - IRCCS Istituti Fisioterapici Ospitalieri, Roma
  - Azienda Ospedaliera Universitaria Senese Policlinico Le Scotte, Siena
- South Korea (7):
  - Kyungpook National University Chilgok Hospital, Daegu, Daegu
  - The Catholic Univ. of Korea, Seoul St. Marys Hospital, Seoul, Seocho-gu
  - Severance Hospital Yonsei University Health System, Seoul, Seodaemun-Gu
  - Samsung Medical Center, Gangam-gu, Seoul
  - Seoul National University Hospital, Jongno-gu, Seoul
  - Asan Medical Center, Songpa-Gu, Seoul
  - Chungnam National University Hospital, Daejeon
- Spain (6):
  - Hospital Universitario Quiron Pozuelo, Madrid, Madrid
  - Hospital Clinic Barcelona, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital General Universitario, Madrid
  - Hospital Regional de Málaga, Málaga
  - Hospital Universitario Miguel Servet, Zaragoza
- Taiwan (3):
  - Taipei Veterans General Hospital, VGHTPE, Taipei, Taipei
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Chang Gung Memorial Hospital LinKou, Taoyuan District
- United Kingdom (3):
  - Royal Marsden Hospital, London
  - The Christie Hospital, Manchester
  - The Churchill Hospital, Oxford

IPD SHARING:
Plan to Share IPD: No